CLINICAL TRIAL: NCT05913752
Title: A Phase I/II Single and Multiple Dose Tolerability, Safety and Pharmacokinetic Study of CMND-100 in Healthy Volunteers and Subjects With Binge Drinking/ Alcohol Use Disorder (AUD)
Brief Title: A First in Human Study of CMND-100 in Healthy and Alcohol Use Disorder (AUD) Subjects
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Clearmind Medicine Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM-CMND-001
Record Dates: First submitted 2023-03-02; First posted 2023-06-22 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: Single and repeated doses of CMND-100. Parts A and B are open-label, non-controlled parts, in which HVs and subjects with binge drinking/AUD respectively will be treated with single, ascending dose cohorts of CMND-100, for evaluation of tolerability, safety and PK/PD. Parts C and D are randomized, double-blind, placebo-controlled parts, in which HVs and subjects with binge drinking/AUD respectively will be treated with repeated doses of CMND-100, for evaluation of safety, PK/PD and preliminary efficacy.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Parts C and D are randomized, double-blind, placebo-controlled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Healthy Subjects - Part A (Other): Part A: Single dose (~ 24 ) Healthy Volunteers: At least four consecutive ascending dose cohorts (20 mg, 40, 80 and 160 mg) will be included in this part of the study in accordance with a pre-defined dose escalating scheme. In each cohort, 6 HVs will receive a single dose of investigation medicine product (CMND-100) starting with the lowest dose of 20 mg. Once dosed, the subjects will be sampled for PK for 24 hours following dosing and will be monitored for drug effects with a physical examination at the end of 24 hours after dosing and daily monitored for safety for a period of 1 week following dosing. Assuming no serious adverse reactions or limiting toxicity (grade 2 and higher) in up to 2, subjects are observed in this dose level, then the next 6 subjects are treated with the next escalated dose, in accordance with a pre-defined dose escalating scheme. The DSMB will review results and guide doses to be studied in Parts B, C and D.
  Interventions: Drug: CMND-100
- AUD Subjects - Part B (Other): Single dose (~12): After DSMB review of part A, binge drinking/AUD subjects will be enrolled in at least 2 consecutive ascending single dose cohorts using the highest tolerable doses from Part A. The first cohort (n=6) will start with the lower ascending dose and sampled for PK for 24 hours following dosing and will be monitored for drug effects with a physical examination at the end of 24 hours after dosing and daily monitored for safety for a period of 1 week following dosing. Assuming no serious adverse reactions or limiting toxicity are observed in this dose level, then the next 6 subjects are treated with the next escalated dose. At the end of this part, real time PK data from the dose cohorts will be collected and analyzed. PK and safety information from this part of the study and from Part A will be reviewed by the DSMB and will guide the dose to be studied in Part D.
  Interventions: Drug: CMND-100
- AUD Subjects - Part C (Placebo Comparator): Multiple dose (18) HVs: Once Part A has been completed, the data analysed and approved by the DSMB, Part C will be initiated. This part will consist of a repeated-dose cohort based on the higher tolerable dose found in Part A. HVs will be randomized into either the treatment or the placebo arm at a ratio of 2:1 (12 subjects treated with the investigation product and 6 subjects receiving placebo) and will receive the drug/placebo at a daily basis for a total of 10 consecutive days. Each subject will be sampled for PK for 24 hours after first and last dosing and will be daily monitored for drug effects and safety throughout the study period and until 1 week after the last dosing. Real time PK data will be collected and results analysed (as defined in Section 5.2). The PK and safety information gathered from in this part of the study will be evaluated by the DSMB and will guide the dose to be studied in Part D of this study.
  Interventions: Drug: CMND-100
- AUD Subjects - Part D (Other): Multiple dose (18) subjects with binge drinking/AUD: Once Part B and Part C has been completed, the data analyzed and approved by the DSMB, Part D will be initiated. This part will consist of a repeated-dose cohort, based on the higher tolerable dose found in Part C and considering the dose effects found in Part B. Subjects will be randomized into either the treatment or the placebo arm at a ratio of 2:1 (12 subjects treated with the investigation product and 6 subjects receiving placebo) and will receive the drug/placebo at a daily basis for a total of 10 consecutive days. Each subject will be sampled for PK for 24 hours after first and last dosing and will be daily monitored for drug effects and safety throughout the study period and until 1 week after the last dosing. The PK and safety information gathered from in this part of the study will be evaluated by the DSMB.
  Interventions: Drug: CMND-100

INTERVENTIONS:
Drug: CMND-100 — The investigational product CMND-100 consists of gelatin capsules, each containing the active ingredient (either 20 or 60 mg) 5-methoxy-2-aminoindane (MEAI) and excipients (stabilizers). MEAI is a psychoactive compound of the aminoindane class
  Other Names: MEAI

SUMMARY:
The primary objective of this study is to find the tolerable dose and characterize the safety and pharmacokinetics/ pharmacodynamics (PK/PD) of single and repeated dose of CMND-100 in Healthy Volunteers (HV) and Subjects with Binge Drinking/Alcohol Use Disorder (AUD).

The secondary objective of this study is to preliminarily evaluate the efficacy of CMND-100 in reduction of drinking patterns and craving in subjects with binge drinking or/and moderate to severe AUD.

DETAILED DESCRIPTION:
This is a Phase I/II, four-parts study (Parts A to D) in HVs and subjects with binge drinking/AUD, evaluating the tolerability, safety, and pharmacokinetics/ pharmacodynamics (PK/PD) of single and repeated doses of CMND-100. Parts A and B are open-label, non-controlled parts, in which HVs and subjects with binge drinking/AUD respectively will be treated with single, ascending dose cohorts of CMND-100, for evaluation of tolerability, safety and PK/PD. Parts C and D are randomized, double-blind, placebo-controlled part, in which HVs and subjects with binge drinking/AUD respectively will be treated with repeated doses of CMND-100, for evaluation of safety, PK/PD and preliminary efficacy. Below is a short description of each part of the study.

* Part A - Single dose (~ 24) HVs: At least four consecutive ascending dose cohorts (20 mg, 40, 80 and 160mg) will be included in this part of the study in accordance with a pre-defined dose escalating scheme (see Section 5.2). In each cohort, 6 HVs will receive a single dose of investigation medicine product (CMND-100) with the first cohort starting with the lowest dose of 20 mg. Once dosed, the subjects will be sampled for PK for 24 hours following dosing and will be monitored for drug effects with a physical examination at the end of 24 hours after dosing and daily monitored for safety for a period of 1 week following dosing. Assuming no serious adverse reactions (as defined in Section 11.1) or limiting toxicity (grade 2 and higher) in up to 2 subjects, as defined in Section 5.2) are observed in this dose level, then the next 6 subjects are treated with the next escalated dose, in accordance with a pre-defined dose escalating scheme. The information gathered in this part of the study will be reviewed by the DSMB and guide the doses to be studied in Parts B, C and D of this study.
* Part B - Single dose (~12) subjects with binge drinking/AUD: Once Part A has been completed and data analyzed and approved by the DSMB, Part B will be initiated and will consist of enrolling subjects with binge drinking/AUD in at least 2 consecutive ascending single dose cohorts using the highest tolerable doses found in Part A. The first cohort will start with the lower ascending dose. Six subjects will be dosed and sampled for PK for 24 hours following dosing and will be monitored for drug effects with a physical examination at the end of 24 hours after dosing and daily monitored for safety for a period of 1 week following dosing. Assuming no serious adverse reactions (as defined in Section 11.1) or limiting toxicity (grade 2 and higher in up to 2 subjects, as defined in Section 5.2) are observed in this dose level, then the next 6 subjects are treated with the next escalated dose. For any grade 2 or higher toxicity in more of two subjects refer to Section 5.2. At the end of this part, real time PK data from the dose cohorts will be collected and analyzed and this information together with the safety information gathered in this part of the study and the data observed in Part A will be reviewed by the DSMB and will guide the dose to be studied in Part D of this study.
* Part C - Multiple dose (18) HVs: Once Part A has been completed, the data analyzed and approved by the DSMB, Part C will be initiated. This part will consist of a repeated-dose cohort based on the higher tolerable dose found in Part A. HVs will be randomized into either the treatment or the placebo arm at a ratio of 2:1 (12 subjects treated with the investigation product and 6 subjects receiving placebo) and will receive the drug/placebo at a daily basis for a total of 10 consecutive days. Each subject will be sampled for PK for 24 hours after first and last dosing and will be daily monitored for drug effects and safety throughout the study period and until 1 week after the last dosing. Real time PK data will be collected, and results analyzed (as defined in Section 5.2). The PK and safety information gathered from in this part of the study will be evaluated by the DSMB and will guide the dose to be studied in Part D of this study.
* Part D - Multiple dose (18) subjects with binge drinking/AUD: Once Part B and Part C has been completed, the data analyzed and approved by the DSMB, Part D will be initiated. This part will consist of a repeated-dose cohort, based on the higher tolerable dose found in Part C and considering the dose effects found in Part B. Subjects will be randomized into either the treatment or the placebo arm at a ratio of 2:1 (12 subjects treated with the investigation product and 6 subjects receiving placebo) and will receive the drug/placebo at a daily basis for a total of 10 consecutive days. Each subject will be sampled for PK for 24 hours after first and last dosing and will be daily monitored for drug effects and safety throughout the study period and until 1 week after the last dosing. The PK and safety information gathered from in this part of the study will be evaluated by the DSMB.

ELIGIBILITY:
Inclusion Criteria:

All Subjects

* Signed informed consent prior to any study-related procedures,
* Subjects understand the nature and the procedures related with the study design of the trial and accept to fulfill all activities related to this trial,
* Subjects 18 to 60 years of age,
* Body mass index between 18 and 35 kg/m2,
* No (history of) clinically significant conditions and/or concomitant medications which in the opinion of the investigator could endanger the safety of the subject or impact the validity of the study results,
* Male subjects who wish use condoms for the duration of the study and for a suitable time period after the last drug dose (e.g., 5 half-lives),
* Female subjects who are not pregnant or breast-feeding or who do not wish to become pregnant during the period of the clinical study and for three months later,
* Female subjects of childbearing potential (less than 24 months after the last menstrual cycle) who use adequate contraceptive methods. Adequate contraceptive methods may include any approved method of birth control such as combined estrogen and progestogen containing hormonal contraception, associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), intra-uterine devices, condoms, abstinence or vasectomized partner. Contraception should be maintained until study end.

Additional Criteria for AUD Subjects

* Non-treatment seeking subjects who report heavy binge drinking (i.e. at least i.e. ≥ 5 standard drinks in a day for men or ≥ 4 standard drinks in a day for women) in at least 5 days in the last month prior to screening OR:
* Treatment seeking subjects with AUD meeting DSM-5 criteria as assessed by SCID and:
* Consumed at least 4 binge drinking days (i.e. ≥ 5 standard drinks in a day for men or ≥ 4 standard drinks in a day for women) in the month prior to screening.
* A desire to reduce or stop drinking.
* Stable housing in the 3 months prior to randomization with no foreseeable risk to lose this in the 3 months after screening,
* Agree to abstain from new/additional psychotropic medications, except for benzodiazepines as rescue medication prescribed by the PI or a stable dose of psychotropic medications in the 1 months prior to randomization with the intention to continue this medication during the study.

Exclusion Criteria All Subjects

* The subject has a clinically significant history of a disease or a disorder that could interfere with the interpretation of the results or could increase the risk to the subject all according to the opinion of the PI.
* Subjects with symptoms of alcohol withdrawal or intoxication at time of screening.
* Subjects with history of seizures or epilepsy,
* Subjects with moderate to severe symptoms of alcohol withdrawal or intoxication at time of screening.
* Subjects positive to HIV at screening,
* Current or past history of Major Depressive Disorder (MDD) (within past 1 years), Bipolar Disorder, Schizophrenia, suicidal ideation (within past 2 years) or suicide attempts in the past 2 years. Individuals suffering from depressed mood who do not meet current criteria for MDD can be included in this trial,
* Uncontrolled inter-current illness (i.e., active infection),
* Clinically significant abnormal vital signs (e.g., systolic blood pressure ≥139 mmHg, diastolic blood pressure ≥90 mmHg, heart rate >90 beats per minute) at separate three measures before dosing,
* Clinically significant abnormal ECG parameters, including subjects with QTc greater than 450 msec,
* Clinically significant abnormal liver functions (ALT and AST), higher than three times the normal amount, clinically significant abnormal Hb,
* Subjects using concomitant medications such as antipsychotic and mood stabilizing medications (including SSRIs such as Fluoxetine and Paroxetine, SNRIs and trazodone), monoamine oxidase inhibitors (MAOIs), tricyclic antidepressants (TCAs), vitamins, herbal and/or mineral supplements, dietary supplements (and/or grapefruit juice), and enzyme altering agents (rifampin, barbiturates, phenothiazines, cimetidine, etc.) or any other medications that may have significant interaction with the study medication, within 2 weeks prior to the study and until the entire duration of study treatment,
* Subjects taking OCT1 and OCT2 substrates,
* Received an experimental drug or used an experimental medical device within 1 month or within a period <5 times the drug's half-life for small molecules, or 3 months for biologics, whichever is longer, before the study drug is administered for the first time,
* Subjects which are in a depression state co-morbidity who take anti depressive drugs on a regular basis,
* Donated blood within 90 days or plasma within 30 days of study dosing,
* Any self-reported current use of drugs such as cocaine, amphetamines, opioids, or barbiturates and/or a positive urine screen for the drugs of abuse just mentioned,
* Any subject who may not be able to fulfill the study requirements per the investigator's clinical judgement.

Additional Criteria for Healthy Subjects

* Subject has a history of drug/substance or alcohol use disorder within 2 years before screening, except for cannabis and nicotine use disorders,
* Subject is unable to abstain from ingesting alcohol for 72 hours prior to dosing.
* Subjects who are symptomatic or requiring ongoing treatment for any mood disorder/event.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Safety as Adverse Events Profile | up to 31 days
  Incidence of adverse events and classification in terms of severity, causality and outcome
Tmax | up to 31 days
  Time to maximum plasma concentration
Cmax | up to 31 days
  Maximum plasma concentration
AUC0-∞ | up to 31 days
  Area under the concentration-time curve from 0 minutes extrapolated to infinity
t1/2 | up to 31 days
  Terminal elimination phase half-life expressed in time units
Cl | up to 31 days
  The volume of plasma cleared of the drug per unit time
Vd | up to 31 days
  The volume in which a drug is distributed

SECONDARY OUTCOMES:
Part D only - Alcohol craving assessment using the Visual Analogue Scale of Craving (VAS) | Change from pre-dose to Day 5 and Days 10 and 17
  VAS was adapted from the Alcohol Craving Questionnaire (ACQ) - Assessment of craving for alcohol based on a 10-point VAS response to the questions "How strong is your craving for alcohol now" where 1 indicates "not at all" and 10 indicates "the most I've ever felt".
Part D only - Assessment of craving for alcohol using the Penn Alcohol Craving Scale (PACS) | The change from pre-dose to Day 5 and Days 10 and 17 of the total score will be evaluated.
  PACS is a questionnaire that includes 5 questions where each question is scored 0 to 6, ranging from the lowest craving-related response (0) to the highest craving-related response (6).

OTHER OUTCOMES:
Assessment of subjective level of sleepiness using the Karolisnka Sleepiness Scale (KSS). (Exploratory Endpoint - 1) | change from pre-dose to Day 5 and Days 10 and 17
  The KSS measures the subjective level of sleepiness at a particular time during the day. On this scale subjects indicate which level best reflects the psycho-physical sate experienced in the last 10 min. The KSS is a 9- point scale (1 = extremely alert, 3 = alert, 5 = neither alert nor sleepy, 7 = sleepy - but no difficulty remaining awake, and 9 = extremely sleepy - fighting sleep).
Assessment of depression symptoms using the Beck Depression Inventory (BDI-II) (Exploratory Endpoint - 2) | The change from pre-dose to Day 5 and Days 10 and 17
  The BDI-II is a widely used, 21- item, self-report measure of depression symptoms. It uses a two-week timeframe to assess the presence of symptoms that include, among others, sadness, guilt, suicidal thoughts, loss of interest, changes in sleep and appetite. Responses are scored from 0 to 3, with 0 representing the absence of the symptom and 4 representing the most severe symptom.
Evaluation of alcohol consumption using Alcohol Timeline Follow-Back (TLFB) (Exploratory Endpoint - 3) | The change from pre-dose to post-dose Day 5 and Days 10 and 17
  TLFB has shown to be a useful tool in the collection of retrospective self-reports of daily alcohol consumption.
Detection of alcohol abuse using alcohol use blood marker gamma-glutamyl transferase (GGT) | The change from pre-dose to post-dose Day 5 and Days 10 and 17
  Increased GGT levels may be detected in the blood before the development of alcohol-related liver injury.
Measurement of chronic alcohol intake using Carbohydrate-deficient transferrin (CDT) | The change from pre-dose to post-dose Day 5 and Days 10 and 17
  CDT has been shown to be an alternative assessment in alcohol abuse patients.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Connecticut Mental Health Center, New Haven, Connecticut
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
- The Sophie and Abram Stuchynski Israeli Alzheimer Medical Center, Ramat Gan, Israel